CLINICAL TRIAL: NCT01220635
Title: Prevention of Depression Within Salient Adolescent Contexts
Brief Title: Middle School Matters Study
Acronym: MSM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Carolyn McCarty, Principal Investigator, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34 MH083706; 5R34MH083076-03 (NIH)
Record Dates: First submitted 2010-10-05; First posted 2010-10-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Depression
Keywords: Depressive Symptoms; Depression prevention; Adolescents; School-Based Services; Health Behavior
MeSH Terms: conditions — Depression; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skill Group Program (Experimental): Positive Thoughts and Actions Program
  Interventions: Behavioral: Positive Thoughts and Actions Program
- Individual Support Program (Active Comparator): Measure of Adolescent Potential for Suicide (MAPS) - modified
  Interventions: Behavioral: Individual Support Program

INTERVENTIONS:
Behavioral: Positive Thoughts and Actions Program — Students in the skills group will attend a 12-session (50 minutes each), 12-week program with 4-6 other students. The skills group will take place at school during school hours. Parents in the skill group will be asked to participate in two parent group workshops to take place at their child's school or other participating middle school (2-hours each). In addition, the skill group leader will conduct two individual family meetings with the student and parent(50 minutes each).
  Arms: Skill Group Program
Behavioral: Individual Support Program — Students will be individually interviewed (60-90 minutes) at school to review areas of stress and support. The health professional conducting the interview will reinforce the student's strengths, and provide connections to sources of help from caring adults at home and at school. Parents will be called following the assessment to help the family locate appropriate resources if needed (e.g., tutoring resources, school counselor).
  Arms: Individual Support Program

SUMMARY:
This study aims to evaluate the short-term and long-term efficacy of two preventative intervention approaches designed to support middle school youth.

DETAILED DESCRIPTION:
This study involve two parts: Part 1 entailed screening 7th and 8th graders from 4 public middle schools to identify students who may be showing moderate signs of stress. Students who score at the designated cutoff on a depression symptoms measure received a brief check-in to determine eligibility for the follow up randomized trial (Part 2). An "indicated" sample of 120 adolescents in the 7th and 8th grade and their caregivers were randomly assigned to a brief, Individual Support Program (ISP) comparison group or a Skills Group Program. Research interviews were conducted at multiple timepoints with students and caregivers, and teacher questionnaires were used to examine changes in outcome measures. Following completion of the intervention, all participants were followed for 12-months.

ELIGIBILITY:
Inclusion Criteria:

* 7th and 8th grade students at 4 participating middle schools
* Score 14 or above on the Mood and Feelings Questionnaire at screening (approximately top 25%)
* No imminent plans to move or change to non-participating school
* At minimum 6th grade language skills
* Agree to participate in random assignment and research interviews
* One Parent/caregiver willing to complete research interviews

Exclusion Criteria:

* Student with past or current Major Depressive Disorder (MDD) or Probable MDD
* Students with parents who do not speak English or Spanish
* Students in concurrent treatment
* Students in self-contained classroom, or with cognitive delays, or emotional behavioral problems that would preclude them from benefiting from the group or being a good group member
* Parent not willing to complete research interviews

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Moods and Feelings Questionnaire (MFQ; child and parent version) | up to 1 year
  Depressive symptoms of the child are assessed on the MFQ. Youth completed the MFQ at all 4 timepoints, parent ratings of students symptoms were collected at baseline, post-intervention, and 12 month follow up.

SECONDARY OUTCOMES:
Parent-Child Communication (PCC; child and parent version) | up to 1 year
  Parent child communication were assessed using the child and parent version of the PCC. Children completed the PCC at all 4 timepoints, parent ratings were collected at baseline, post-intervention, and 12 month follow up.
Behavioral Assessment System for Children-2nd Edition (BASC-2; student, parent, & teacher version) | up to 1 year
  The adolescent version of the Teacher Rating Scale, Parent Rating Scale, and the Student Self-Report of Personality of the BASC-2 were used to assess school functioning and social functioning.
Health Enhancing Behavior Index (HEBI) | up to 1 year
  Health behaviors (diet, exercise, and sleep) are self-reported by the youth on the HEBI.
Service Use Interview (Service for Children and Adolescence Parent Interview-modified) | up to 1 year
  The service use interview was used to measure treatment history and services received during the course of the intervention and follow up.
Schedule for Affective Disorders and Schizophrenia for School-Age Children (KSADS) | up to 1 year
  The depression module of the KSADS was used to assess DSM-IV symptoms of major depression and depressive disorder at the 12-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn A McCarty, Ph.D., Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's, Seattle, Washington, United States

REFERENCES:
- [Derived] Duong MT, Kelly BM, Haaland WL, Matsumiya B, Huey SJ Jr, McCarty CA. Mediators and Moderators of a School-Based Cognitive-Behavioral Depression Prevention Program. Cognit Ther Res. 2016 Oct;40(5):705-716. doi: 10.1007/s10608-016-9780-2. Epub 2016 Apr 28. PMID 27795599